CLINICAL TRIAL: NCT06903767
Title: Do Quantifiable Differences in Physiologic Stress Exist in Surgeons When Comparing the Use of a Powered Femoral Impactor Versus Manual Impaction in Total Hip Arthroplasty?
Brief Title: Automated V Manual Impactor Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: UCLA Health - Santa Monica Medical Center (Unknown); University of Virginia (Other); Orthopedic + Fracture Specialists, Portland, OR (Other)
Responsible Party: Principal Investigator, tnicholson, Director of Clinical Trials, Rothman Institute Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JLON1384286
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Total Hip Arthroplasty (THA); Impaction; Physiological Strain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Manual Malleting Group (Active Comparator): For cases that are randomized to the manual malleting group, surgeons will utilize a manual mallet to perform impaction during total hip arthroplasty while wearing the Hexoskin shirt.
  Interventions: Device: Manual Malleting
- Automated Impaction HAMMR Group (Active Comparator): For cases that are randomized to the automated impaction HAMMR group, surgeons will utilize an automated impaction device to perform impaction during total hip arthroplasty while wearing the Hexoskin shirt.
  Interventions: Device: Automated Impaction (HAMMR)

INTERVENTIONS:
Device: Automated Impaction (HAMMR) — For cases that are randomized to the automated impaction HAMMR group, the surgeon will utilize an automated impactor device for impaction of the implant during total hip arthroplasty.
  Arms: Automated Impaction HAMMR Group
Device: Manual Malleting — For cases that are randomized to the manual malleting group, the surgeon will utilize a mallet for impaction of the implant during total hip arthroplasty.
  Arms: Manual Malleting Group

SUMMARY:
This study investigates the use of an automated impactor device in total hip arthroplasty versus manual malleting method and the physiological strain on the surgeon. This study will be a randomized, prospective, multicenter study involving fellowship-trained arthroplasty surgeons. Each participating surgeon will contribute data from 50 primary, elective THA cases, using the HAMMR powered impactor in 25 cases and manual impaction in 25 cases.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing primary elective THAs Participants over the age of 18 Patients with compatible implants

Exclusion Criteria:

Attending orthopaedic surgeons with pre-existing cardiorespiratory or musculoskeletal conditions Use of cemented or hybrid THA Patients undergoing a conversion or revision THA Patients undergoing a non-elective THA (i.e., for fracture) Participants lacking cognitive capacity to consent Participants who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Physiological strain in the surgeon | 1 day
  Through the use of a Hexoskin vest worn by the surgeon, we will measure heart rate, heart rate variability, respiratory rate, minute ventilation, and energy expenditure to determine overall physiological strain on the surgeon during total hip arthroplasty.

SECONDARY OUTCOMES:
Patient Adverse Events | 6 weeks
  Patient adverse events such as periprosthetic fractures intra- or postoperatively, intraoperative soft tissue injury, etc. will be recorded intra or postoperatively.
F-NRS | 1 day
  We will assess the Fatigue numeric rating scale (F-NRS) of surgeons after each case via survey.

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Restrepo, MD, Study Director — Rothman Orthopaedic Institute
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States